CLINICAL TRIAL: NCT04752007
Title: Accuracy of the CT-Implant Movement Analysis. A Feasibility Study.
Brief Title: Movement of the Sacroiliac (SI) Joint, Comparing Conventional RSA With the Sectra Implant Movement Analysis.
Acronym: IMSRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IMSRA
Record Dates: First submitted 2020-10-27; First posted 2021-02-12 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Sacroiliac Instability
MeSH Terms: interventions — Supine Position

STUDY DESIGN:
Intervention Model Description: One group will be measured using conventional RSA and the other using low dose CT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RSA group (Active Comparator): Conventional RSA to measure the movement in th SI joint.
  Interventions: Radiation: ASLR; RSA; SI joint movement: stright leg raise with 1 kg load; Radiation: Fig.Four; RSA; SI joint movement: One side figure of four position with 1 kg load; Radiation: Supine; RSA; SI joint movement: supine position
- CT group (Active Comparator): Low dose CT to measure the movement in th SI joint.
  Interventions: Radiation: ASLR; CT; SI joint movement: stright leg raise with 1 kg load; Radiation: Fig.Four; CT; SI joint movement: One side figure of four position with 1 kg load; Radiation: Supine; CT; SI joint movement: supine position

INTERVENTIONS:
Radiation: ASLR; CT; SI joint movement: stright leg raise with 1 kg load — Measurement of the SI joint movement in mikrometer
  Arms: CT group
Radiation: Fig.Four; CT; SI joint movement: One side figure of four position with 1 kg load — Measurement of the SI joint movement in mikrometer
  Arms: CT group
Radiation: Supine; CT; SI joint movement: supine position — Baseline position
  Arms: CT group
Radiation: ASLR; RSA; SI joint movement: stright leg raise with 1 kg load — Measurement of the SI joint movement in mikrometer
  Arms: RSA group
Radiation: Fig.Four; RSA; SI joint movement: One side figure of four position with 1 kg load — Measurement of the SI joint movement in mikrometer
  Arms: RSA group
Radiation: Supine; RSA; SI joint movement: supine position — Baseline position
  Arms: RSA group

SUMMARY:
Movement of the Sacroiliac (SI) Joint, comparing conventional RSA with the Sectra Implant Movement analysis using a low dose CT for high accuracy measurement. A feasibility study for a future kohort study.

DETAILED DESCRIPTION:
Abstract Background: Radiostereometric analysis (RSA) is a high precision in vivo measuring method and regarded as the gold standard for motion analysis. RSA has been around for over 40 years and its accuracy is properly evaluated. The CT technics have evolved and now low dose CT scans can reproduce 3-D models of bone and joints. The Sectra Implant Movement analysis (IMA) is a new method using a low dose CT for high accuracy measurement. There is no study evaluating the precision and accuracy of the new CT based method.The investigator want to compare the accuracy of the two methods.

Method/design: The RSA method will be tested in patients that already have tantalum markers inserted around the SI joints from earlier studies conducted at Ullevål University Hospital. There are 2-6 patients in the age of 40-50 years available for RSA analysis with and without provocation of the SI joints. Some are fused in one SI joint after insertion of the tantalum markers, but the contralateral joint can then be used for the analysis. At the same time,the investigator will perform low dose CT with and without provocation of the SI joints. The results of the analysis will be compared.

Discussion: The conventional RSA is an invasive method using tantalum markers inserted in to bone. If the CT method has the same accuracy, then the tantalum markers will become obsolete and future studies can easily be performed using non-invasive low dose CT scans.

Keywords: RSA, CT method, low dose CT, IS joint, movement

Introduction:

Because of the high accuracy and precision, radiostereometric analysis (RSA), has become a well- established method for three-dimensional (3-D) measurements of micro motion in joints. The implantation of tantalum markers is invasive, but no reports of patient injuries are reported. The markers might be inserted through the approach used during a surgical intervention or in an extra stab incisions in the skin to get the markers to the necessary position in the bony structures. The placements of the markers are of outmost importance to achieve good quality measurements. At least three no collinear markers in each segment and a good distance and distribution in all three axes (X, Z, Y) is essential for a good 3-D configuration.

The CT techniques have evolved and now low dose CT scans can reproduce 3-D models of bone and joints. The Sectra Implant movement analysis (IMA) is a non-invasive method using a low dose CT scan. No tantalum markers are needed and joint provocation can easily be conducted in the CT. The CT scan is then sent to the Sectra AB for analysis.

Method:

Patients and methods:

The RSA method will be tested in patients that already have tantalum markers inserted around the SI joints from earlier studies , approximately five years ago, conducted at Ullevål University Hospital. These are patients with long lasting severe sacroiliac joint pain. There are six patients in the age of 40-50 years available for RSA analysis with and without provocation of the SI joints, at the same time the investigator will perform low dose CT with and without provocation of the SI joints. For the non-provocation, the patient will be in a supine-position. The provocation x-ray/low dose CT will be performed; 1: anterior straight leg raise 2: One side figure of four position, both with 1kg of load. Some are fused in one SI joint after insertion of the tantalum markers, but the contralateral joint can then be used for the analysis. The investigators will also measure eventual movement in the fused joint and the symphysis (if tantalum markers present). The Center for Implant and Radiostereometric Research Oslo has extensive experience with RSA and established state of the art measuring method of movement in the SI joint. They will perform the RSA measurements. The CT scan is send to the Sectra AB for analysis.

Statistical analysis:

Null hypothesis (H0): There is no difference in the accuracy Alternate Hypothesis (H1): There is a difference in the accuracy Continuous variables will be described with mean and standard deviation\, and the normality of the data will be checked using the histograms, QQ-plots and the Kolmogorov-Smirnov-Test of normality. The differences of motion will also be tested for normality. The paired sample T-test will be used to detect possible significance in the difference between the two groups. Non-parametric tests are used if the assumption of normality does not hold. All analysis will be conducted using commercially available software (SPSS version 24, IBM Inc.) and the level of significance is set to p<0.05 in a two-sided test.

Participants Project leader and responsible institution Stephan M. Röhrl, PhD, MD, Ass. Professor, Head of Center for Implant and Radiostereometric Research Oslo, President of Knee and Hip Register, Oslo University Hospital, Oslo, Norway.

PhD candidate Vinjar Myklevoll, MD, Haukeland University Hospital, Bergen. Collaborating partner Thomas Kibsgård, Ass. Professor, PhD, MD, President Pelvic Girdle Pain Society, Head of Department Rikshospitalet, Oslo, OUS.

ELIGIBILITY:
Inclusion Criteria:

* The RSA method will be tested in patients that already have tantalum markers inserted around the SI joints from earlier studies, approximately five years ago, conducted at Ullevål University Hospital.

Exclusion Criteria:

* The patients that can not perfome the provocation images of the SI joints.
* Pregnancy
* Not able to or do not want to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Movement of the SI joint in mikrometer | 4 weeks
  Movement analysis

CONTACTS AND LOCATIONS:
Overall Officials: Stephan M Rohrl, PhD, Study Director — Oslo University Hospital
Locations (1):
- Cirro at Ullevål Uiversity Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
There are only two researchers in the study, Stephan M. Röhrl and Vinjar Brenna Hansen. The participant data will only be available for them.

REFERENCES:
- [Background] Axelsson P, Karlsson BS. Intervertebral mobility in the progressive degenerative process. A radiostereometric analysis. Eur Spine J. 2004 Oct;13(6):567-72. doi: 10.1007/s00586-004-0713-5. Epub 2004 May 19. PMID 15150701
- [Background] Fayyazi AH, Ordway NR, Park SA, Fredrickson BE, Yonemura K, Yuan HA. Radiostereometric analysis of postoperative motion after application of dynesys dynamic posterior stabilization system for treatment of degenerative spondylolisthesis. J Spinal Disord Tech. 2010 Jun;23(4):236-41. doi: 10.1097/BSD.0b013e3181a4bb0b. PMID 20072031
- [Background] Nabhan A, Al-Yhary A, Ishak B, Steudel WI, Kollmar O, Steimer O. Analysis of spinal kinematics following implantation of lumbar spine disc prostheses versus fusion: radiological study. J Long Term Eff Med Implants. 2007;17(3):207-16. doi: 10.1615/jlongtermeffmedimplants.v17.i3.40. PMID 19023945
- [Background] Sturesson B, Uden A, Vleeming A. A radiostereometric analysis of the movements of the sacroiliac joints in the reciprocal straddle position. Spine (Phila Pa 1976). 2000 Jan 15;25(2):214-7. doi: 10.1097/00007632-200001150-00012. PMID 10685486
- [Background] Sturesson B, Uden A, Vleeming A. A radiostereometric analysis of movements of the sacroiliac joints during the standing hip flexion test. Spine (Phila Pa 1976). 2000 Feb 1;25(3):364-8. doi: 10.1097/00007632-200002010-00018. PMID 10703111
- [Background] Zoega B, Karrholm J, Lind B. Plate fixation adds stability to two-level anterior fusion in the cervical spine: a randomized study using radiostereometry. Eur Spine J. 1998;7(4):302-7. doi: 10.1007/s005860050079. PMID 9765038
- [Background] Broden C, Olivecrona H, Maguire GQ Jr, Noz ME, Zeleznik MP, Skoldenberg O. Accuracy and Precision of Three-Dimensional Low Dose CT Compared to Standard RSA in Acetabular Cups: An Experimental Study. Biomed Res Int. 2016;2016:5909741. doi: 10.1155/2016/5909741. Epub 2016 Jul 10. PMID 27478832
- [Background] Broden C, Sandberg O, Skoldenberg O, Stigbrand H, Hanni M, Giles JW, Emery R, Lazarinis S, Nystrom A, Olivecrona H. Low-dose CT-based implant motion analysis is a precise tool for early migration measurements of hip cups: a clinical study of 24 patients. Acta Orthop. 2020 Jun;91(3):260-265. doi: 10.1080/17453674.2020.1725345. Epub 2020 Feb 14. PMID 32056507
- [Background] Nagamoto Y, Iwasaki M, Sakaura H, Sugiura T, Fujimori T, Matsuo Y, Kashii M, Murase T, Yoshikawa H, Sugamoto K. Sacroiliac joint motion in patients with degenerative lumbar spine disorders. J Neurosurg Spine. 2015 Aug;23(2):209-16. doi: 10.3171/2014.12.SPINE14590. Epub 2015 May 15. PMID 25978076
- [Background] Forsth P, Svedmark P, Noz ME, Maguire GQ Jr, Zeleznik MP, Sanden B. Motion Analysis in Lumbar Spinal Stenosis With Degenerative Spondylolisthesis: A Feasibility Study of the 3DCT Technique Comparing Laminectomy Versus Bilateral Laminotomy. Clin Spine Surg. 2018 Oct;31(8):E397-E402. doi: 10.1097/BSD.0000000000000677. PMID 29939843
- [Background] Svedmark P, Berg S, Noz ME, Maguire GQ Jr, Zeleznik MP, Weidenhielm L, Nemeth G, Olivecrona H. A New CT Method for Assessing 3D Movements in Lumbar Facet Joints and Vertebrae in Patients before and after TDR. Biomed Res Int. 2015;2015:260703. doi: 10.1155/2015/260703. Epub 2015 Oct 26. PMID 26587533
- [Background] Svedmark P, Tullberg T, Noz ME, Maguire GQ Jr, Zeleznik MP, Weidenhielm L, Nemeth G, Olivecrona H. Three-dimensional movements of the lumbar spine facet joints and segmental movements: in vivo examinations of normal subjects with a new non-invasive method. Eur Spine J. 2012 Apr;21(4):599-605. doi: 10.1007/s00586-011-1988-y. Epub 2011 Sep 1. PMID 21881866
- [Background] Eriksson T, Maguire GQ Jr, Noz ME, Zeleznik MP, Olivecrona H, Shalabi A, Hanni M. Are low-dose CT scans a satisfactory substitute for stereoradiographs for migration studies? A preclinical test of low-dose CT scanning protocols and their application in a pilot patient. Acta Radiol. 2019 Dec;60(12):1643-1652. doi: 10.1177/0284185119844166. Epub 2019 May 1. No abstract available. PMID 31042065
- [Background] Kibsgard TJ, Rohrl SM, Roise O, Sturesson B, Stuge B. Movement of the sacroiliac joint during the Active Straight Leg Raise test in patients with long-lasting severe sacroiliac joint pain. Clin Biomech (Bristol). 2017 Aug;47:40-45. doi: 10.1016/j.clinbiomech.2017.05.014. Epub 2017 May 29. PMID 28582642
- [Background] Kibsgard TJ, Roise O, Stuge B, Rohrl SM. Precision and accuracy measurement of radiostereometric analysis applied to movement of the sacroiliac joint. Clin Orthop Relat Res. 2012 Nov;470(11):3187-94. doi: 10.1007/s11999-012-2413-5. Epub 2012 Jun 14. PMID 22695864

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT04752007/Prot_SAP_000.pdf